CLINICAL TRIAL: NCT01202136
Title: The Clinical,Radiologic, Pathologic and Molecular Marker Characteristics of Premalignant and Malignant Pancreatic Cysts Study
Brief Title: The Clinical,Radiologic,Pathologic and Molecular Marker Characteristics of Pancreatic Cysts Study
Acronym: PCyst
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Lustgarten Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00026447
Record Dates: First submitted 2010-09-09; First posted 2010-09-15 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cysts; Pancreatic Cancer
Keywords: pancreatic cyst; IPMN; PAN INs; Pancreatic cancer; pancreatic neoplasia
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, pancreatic cyst fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic cysts: patients referred to Johns Hopkins Hospital for evaluation and or treatment for 1 or more pancreatic cysts

SUMMARY:
The aim is to propose and prospectively validate a diagnostic approach and model for prediction of mucinous versus non-mucinous, and malignant versus non-malignant pancreatic cysts using a combination of clinical, radiologic, and biomarker characteristics.

DETAILED DESCRIPTION:
This combined cross-sectional and prospective single center clinical and translational study involves a collaborative multidisciplinary team composed of gastroenterologists, surgeons, radiologists, and basic scientists. Eligible patients with solitary or multiple pancreatic cysts referred for diagnostic evaluation and/or surgical treatment will undergo initial radiographic imaging with high-resolution CT, MRI/MRCP, and EUS/FNA as part of standard medical care at Johns Hopkins Hospital. This is a three-phase study.

In Phase I, eligible patients with pancreatic cysts will undergo initial radiographic imaging (high-resolution CT, MRI/MRCP, endoscopic ultrasonography (EUS) with fine needle aspiration (FNA)) as part of standard care at the Johns Hopkins Hospital. Patients will be categorized according to the presence of symptoms referable to the cyst or imaging features concerning for malignancy based on the initial radiographic assessment. Symptomatic patients, or those with concerning features, will be referred for surgical resection. The pathologic features and final diagnosis of resected pancreatic cysts will be compared with preoperative clinical, radiologic, and cyst fluid test results.

Asymptomatic patients with low-risk features at baseline radiographic and endoscopic imaging will enter Phase II. Patients will be followed on a prospective periodic surveillance schedule according the consensus clinical guidelines with either CT or MRI to monitor for new or metachronous cystic neoplasms. Those who develop symptoms or concerning features will have a repeat EUS/FNA as well as imaging with the opposite axial imaging modality, and will be referred for surgery if a suspicious lesion is detected.

Patients who have surgery either during Phase I or Phase II, will enter post-surgical surveillance (Phase III). Patients will be followed using a prospective periodic surveillance schedule according the consensus clinical guidelines with either CT or MRI to monitor for new or metachronous cystic neoplasms. Those who undergo surgery after surveillance in Phase II will continue with the imaging modality they were originally evaluated with prior to surgery.. Patients who develop symptoms or high-risk features on imaging will have a repeat EUS/FNA as well as imaging with the opposite axial imaging modality and will be referred for surgery if a suspicious lesion is detected. Samples will be collected prospectively for biomarker analysis. Cyst fluid, pancreatic juice and blood will be collected during EUS and blood will be collected yearly during the outpatient clinic visit. Patients will be followed for three years.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age 18 years and older
2. Referred for assessment of one or more pancreatic cyst.

Exclusion Criteria:

1. Medically ill patients with ASA class 4 or greater.
2. History of chronic kidney disease with a serum creatinine > 2.0 mg/dl or estimated glomerulofiltration rate (eGFR) < 30 ml/min, dialysis patients, acute renal failure, cirrhosis of the liver, chronic hepatitis, prior nephrectomy or kidney or liver transplantation.
3. History of moderate (generalized hives) or severe (facial swelling, airway reaction) reaction to intravenous radiographic contrast material.
4. History of obstruction in the upper GI tract such as esophageal or pyloric stricture, which would not allow passage of an endoscope.
5. Bleeding diathesis (clotting problems) or a history of thrombocytopenia (low platelet count <50,000).
6. Inability to provide informed consent.
7. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to Johns Hopkins for evaluation of pancreatic cysts
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2012-10; Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Prevalence and incidence of malignant pancreatic cysts | 3-6 years
  1)to determine the prevalence and incidence of malignancy in pancreatic cysts according to cyst size and concerning features

SECONDARY OUTCOMES:
Biomarkers to predict type of pancreatic cyst | 3-6 years
  To collect tissue samples (cyst fluid and blood) for research on molecular markers in pancreatic cysts
Biomarker panel in pancreatic juice as indicator to type of pancreatic cyst | 3-6 years
  To develop a panel of candidate biomarkers in pancreatic juice and serum as indicators of prevalent and incident malignancy in patients with surgically-proven neoplastic pancreatic cysts compared to non-neoplastic cysts (pseudocysts, lymphoepithelial cysts, congenital cysts)
Compare CT with EUS and MRI for diagnosing pancreatic cysts. | 3-6 year
  to determine the sensitivity, specificity, and overall accuracy of pancreatic protocol CT, EUS, and/or MRCP in patients with pancreatic cysts, using surgical pathology as the reference standard
Difference EUS/CT or MRCP in diagnosis of malignant pancreatic cysts | 3-6 years
  to calculate difference in diagnostic accuracy and clinical impact (change in preoperative diagnosis and treatment plan) of additional diagnostic tests (EUS and/or MRCP) over pancreatic protocol CT for the diagnosis of neoplastic/malignant pancreatic cysts.
Associated factors for with multivariate model for malignant pancreatic cyst | 3-6 years
  to determine the factors associated with prevalent and incident malignancy in pancreatic cyst using a multivariate model including clinical, radiologic, and molecular markers
Model for prediction of malignant pancreatic cysts | 3-6 years
  to determine the best model for prediction of malignancy in pancreatic cysts using multiple logistic regression and discriminant function analysis, including clinical, radiologic, and molecular markers

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie O'Broin-Lennon, MD, Principal Investigator — John Hopkins University, School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Medicine, Baltimore, Maryland